CLINICAL TRIAL: NCT05159167
Title: Impact of Baduanjin Qigong Exercise on Fatigue in Patients With Non Small Cell Lung Cancer Undergoing Adjuvant Chemotherapy: A Randomized Controlled Trial
Brief Title: Impact of Baduanjin Qigong Exercise on Fatigue in Patients With NSCLC Undergoing Adjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yu Qian, Doctor, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LLHBCH2021YN-029
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group received two months of Baduanjin exercise training provided by the specialist coach 3 days per week in Hubei Cancer Hospital, and they were also required to do Baduanjin exercise at home for the remaining 4 days each week for at least 20 min per day. All the participants are requested to monitor and record adverse effects during their exercise sessions.
  Interventions: Other: Baduanjin, a type of Qigong
- Control group (Placebo Comparator): Participants in the control group were requested to maintain their original daily physical activity for no less than 20 min per day over the following 6-month period and record their daily activity at home by themselves. These data were collected by a researcher during the participants' time in the study and at the 6-month follow-up at the hospital. After the 6-month follow-up, the participants were provided with 1-month professional Baduanjin exercise guidance by the trial's specialist coach for free if they wished.
  Interventions: Other: Baduanjin, a type of Qigong

INTERVENTIONS:
Other: Baduanjin, a type of Qigong — Baduanjin is very popular in China. There is increasing evidence to support its positive effects on health outcomes in various groups of people with physical and mental disorders.

SUMMARY:
Baduanjin，a type of Qigong which belongs to aerobic exercise, is very popular in China. There is increasing evidence to support its positive effects on health outcomes in various groups of people with physical and mental disorders. In college students, it may enhance cardio respiratory function, lower limb function, and flexibility compared with usual exercise. However, there is no previous relevant randomized controlled trials on the health promoting effects of Baduanjin exercise in targeted fatigued lung cancer patients. Lung cancer survivors can experience fatigue due to multiple reasons that can strongly impact their quality of life throughout the remainder of their life. Therefore, this randomized controlled trial in China was designed to assess the health promoting effects of Baduanjin exercise in fatigued lung cancer patients with the expectation of improvement in physical and psychological health.

ELIGIBILITY:
Inclusion Criteria:

* This trial aims to enroll 18- to 75-year-old patients expected to survive > 3 months and with a Zubrod performance status of 0 to 2. All patients must have diagnosed as lung cancer and have at least one cycle of adjuvant chemotherapy. Enrolled patients should have a minimal ESAS fatigue as 3. Other inclusion criteria are lack of leptomeningeal disease, adequate hepatorenal function and blood counts (red blood cells, >3.0 * 1012/L; white blood cells, > 3.5 * 109/L; absolute neutrophil count, > 1.5 * 109/L; platelets, > 100 * 109/L; hemoglobin > 90 g/L).

Exclusion Criteria:

* Children

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Scale of fatigue | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wu, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided